CLINICAL TRIAL: NCT02403752
Title: Paired Integrative Home Exercise for Seniors With Dementia and Their Caregivers
Brief Title: Paired Integrative Home Exercise for Seniors With Dementia and Their Caregivers (PairedPLIE)
Acronym: PairedPLIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-14943
Record Dates: First submitted 2015-03-18; First posted 2015-03-31 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Dementia; Alzheimer's Disease
Keywords: dementia; Alzheimer's disease; exercise
MeSH Terms: conditions — Dementia; Alzheimer Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- exercise intervention (Experimental): Exercise protocol based on the PLIÉ protocol, developed in consultation with experts worldwide, incl. traditional strength-building exercises, yoga, Tai Chi and Feldenkrais, that engage the muscles most needed to maintain independence--including lower body strength, balance, upper body strength, fine motor exercises , and pelvic floor exercises- combined them into a unique integrative exercise program, to be purposeful and to build procedural ('muscle') memory.
  To be practiced at home in dyads of affected individuals and caregivers, called Paired PLIE Program.
  Interventions: Behavioral: Paired PLIE Program

INTERVENTIONS:
Behavioral: Paired PLIE Program — Integrative exercise as described above

SUMMARY:
Specific Aim 1: To determine feasibility of a 20-minute dyadic exercise program for ambulatory individuals with dementia and caregivers living at home based on recruitment, adherence and retention. Investigators will conduct a pilot randomized controlled trial (RCT) with 20 dyads (total N = 40) in groups of 5 randomized to 16-week group exercise classes and regular home practice or wait list in a cross-over design. Investigators will assess feasibility of enrollment and retention, the proportion of completed outcome measures, and adherence by class attendance logs, caregiver-reported home practice logs and qualitative interviews to assess ease of implementation in the home environment. Investigators will explore feasibility of weekly phone calls to (potentially overwhelmed) caregivers and Fit-bit accelerometers as a measure for tracking home practice.

Specific Aim 2: To collect preliminary effect size data for sample size calculation for a larger trial. Investigators will assess standard outcomes (such as the Short Physical Performance Battery and Alzheimer's Disease Assessment Scale - cognitive subscale as primary outcomes for affected individuals; and Caregiver Burden Inventory for caregivers) commonly used in pharmacological studies of individuals with dementia at baseline, 16 and 32 weeks and calculate effect sizes (Cohen's d) for between-group differences in outcome changes in the 20 dyads of the RCT described in Specific Aim 1.

Specific Aim 3: To explore the feasibility of using non-invasive Near-Infrared Spectroscopy (NIRS) to assess regional cortical brain oxygenation and its sensitivity to change. Investigators will compare brain oxygenation variations before and after the exercise intervention during a memory task for the seniors with dementia.

DETAILED DESCRIPTION:
Alzheimer's dementia (AD) is a major public health challenge for our century. Research into pharmaceutical therapies has been disappointing and not provided any safe medications that can halt the disease's trajectory of decline in the cognitive, functional, emotional and social capabilities of the affected individuals. For non-pharmacological approaches, multi-domain exercise programs that address several of these capabilities in an integrated way have shown strong promise for their ability to slow the decline. The team of investigators has systematically developed one such program-the Preventing Loss of Independence through Exercise (PLIÉ) program-an integrative exercise program that uses procedural memory (memory for movements without explicit recall), can be taught at and integrated into senior day care centers and has been pilot-tested by our team with encouraging results for functional, cognitive and social outcomes (see Table 1).

However, (1) most people in the community do not have access to a day care center, are concerned about the stigma associated with day care or are unable to afford it. This was endorsed by semi-structured interviews conducted with caregivers and community-based organizations in preparation for a larger study of the PLIÉ program. There is a huge need for innovative programs to assist individuals with dementia and their caregivers in the community. Irrespective of having access to day care or not, motivated caregivers, who are aware of the benefits of exercises for their loved ones and spend hours alone with them at home, ask: "What can we do with our [e.g. mother]?" They point out a major lack of guidance for caregivers in the community to be able to use a regular exercise practice on a long-term basis at home. Caregivers and seniors with dementia living together in the community are dyads in need of a paired exercise program. (2) How exercise may delay cognitive and functional decline is unknown. One hypothetical mechanism of action is an improved brain oxygenation related to exercise. Near-Infrared Spectroscopy (NIRS) is a non-invasive method to assess regional cortical oxygenation levels, has been suggested for the early diagnosis of Alzheimer's dementia, but has never been applied to longitudinal studies in this population.

Paired home exercise programs for seniors with dementia and their primary caregivers have rarely been studied. A pilot study that used 6 'sticky hands' movement variations based on Tai Chi, music and exercise incentives found improvements in 2 outcome measures considered to be important in fall prevention (sit-to-stand time, one-legged stance time). However, movements were limited to tai chi and outcomes to fall-related function, leaving out cognitive function for which the PLIÉ program had shown such promising results.

The group of investigators is an established collaboration between the Osher Center for Integrative Medicine and the Department of Psychiatry at UCSF and has recently pioneered a novel, 45-minute, multi-domain program called Preventing Loss of Independence through Exercise (PLIÉ) that integrates physical activity (training of procedural memory for basic daily activities such as sitting and standing), cognitive stimulation (mindful body awareness), social engagement (group movement and sharing of in-the-moment experiences), and caregiver education (monthly home-visit). The investigators pilot-tested PLIÉ in 11 individuals with mild to moderate dementia who were attending an adult day program at the Institute of Aging in San Francisco, CA (ClinicalTrials.gov registered NCT01371214), and found (Table 1) preliminary evidence of medium to large, clinically meaningful effect sizes com-pared to usual care (UC; 45 minutes of usual chair-based exercises at the day care center) across a wide range of out-comes including measures of quality of life (0.83), cognitive function (0.76), physical performance (0.34) and caregiver burden (0.49).7,11 That study methodologically mimicked a drug study by including measures that are commonly used in dementia medication trials, which enabled comparison of the magnitude of our results to currently available dementia medications.. The investigators are now completing data collection for a second implementation of the PLIÉ program at an adult day program in San Rafael, CA (Senior Access). The intervention of the current proposal will be similar to PLIÉ in using the same principles6 and taught by instructors trained in the PLIÉ program. However, it will differ in its format: instead of a day-care center-based group program taught by professional exercise instructors, it uses a dyadic approach, introduced through caregiver support groups to pairs of individuals with dementia and their caregivers, initially using a group class format, but taught to enable caregivers to practice independently at home. To allow for wide-spread long-term routine application, it will be brief (20 minutes), use personalized music associated with positive affect memories, and be supported by video instructions.

2 papers have been published about the study.

Therefore, the investigators propose studying a paired integrative exercise intervention that can be practiced in dyads of caregivers and affected individuals at home or in a community-based support group environment, does not require additional equipment, can be easily learned by caregivers, and may ameliorate the impact of dementia for older persons and caregivers. The investigators suggest a multimodal program that is based on implicit procedural learning and the integrative principles of the PLIÉ program: it includes physical (through touch) and social interaction with a trusted family member, focuses on physical function such as balance, includes personalized music choices and singing, supports positive affect, and uses language to cognitively enhance the experience of mind-body integration. It promotes a playful, non-judgmental supportive attitude to foster a sense of embodied personhood in individuals with dementia through joyful social interaction with an empowered caregiver.

1. Recruitment. Study participants will be recruited from local caregiver support groups of Kaiser Permanente in Oakland. Exercise instructors and the PI have already been invited to give presentations at their regular meetings. Contacts have been established with 3 caregiver support groups meeting at Kaiser Permanente in Oakland, totaling about 100 caregivers, who meet once a month and confirmed strong interest to participate. Thus, it is highly likely that we will twice be able to recruit 10 dyads of eligible participants. In addition, investigators will give study flyers to caregiver support managers at Kaiser Permanente, the local Alzheimer's Association groups, and the Alzheimer's Services of the East Bay (ASEB). In addition, we will recruit at ASEB.

   Caregivers will be informed about the study by brief presentations by the PI and an exercise instructor during regular support group meetings. A flyer will be handed to interested potential participants describing the study and providing an opportunity to learn more by returning a form or calling the research study staff. Those caregivers who express interest will be contacted by research staff by phone to further assess interest/eligibility and to schedule a consent visit.
2. Informed consent. Verbal consent to be screened will be obtained over the telephone prior to collecting information on demographics and medical and psychiatric history. Written consent will be obtained with the affected individuals and caregivers together, as described in more detail below. The consent forms will be reviewed and capacity to consent will be assessed in primary participants based on responses to questions to determine level of understanding of study procedures, risks, benefits and rights. Participants who do not demonstrate capacity to consent will be asked to assent to study procedures and caregivers will be asked to consent on their behalf. A separate consent form will request permission to participate in video recording of exercise classes for quality control purposes. After the consent process has been completed, the Modified Mini-Mental State Exam (3MS) will be administered to affected individuals to assess level of cognitive impairment. Consent procedures will take place at the Kaiser group room unless otherwise requested by caregivers.

   If the caregiver is not the Legally Authorized Representative (LAR) or the legal guardian of the affected individual, the screening interview will be stopped. Investigators will then mail a letter to the LAR or legal guardian and invite her/him to contact us by mail or phone to discuss the study and the consent process. The screening and eligibility questions for the affected individual will then be completed with the LAR or legal guardian. If investigators do not get a response within 2 weeks they will call the LAR or legal guardian by phone assuming that she/he has received our letter. Only if this person permits the affected individual's study participation investigators will contact the caregiver and the affected individual again.

   How will investigators assess the potential participant's capacity to consent? Capacity to consent will be assessed by research assistants (RA) who will be extensively trained by the PI and co-investigators using a standardized procedure. Investigators first provide the consent form to the patient and caregiver together and allow them to review it. RAs then describe the key points of the form, pointing to the areas on the form where the information is described in more detail. They then ask a series of yes/no questions to assess understanding of the information in the form. If the participant cannot answer the questions, RAs review the material again and point to the section on the form. Investigators then repeat the questions. If participants are unable to answer all of the questions on their own after review, RAs consider them to lack capacity to consent. RAs then ask them if they would like to participate in the study to obtain their assent. RAs say that they are going to ask the caregiver to sign the form on the participant's behalf to obtain written consent. Most of the team's research assistants have been and are psychology graduate students who are highly sensitive to working with vulnerable patients. Investigators train new research staff by having them role play the consent process until senior personnel determine that they are adequately prepared. They then observe senior personnel performing the consent process on at least one study participant. Subsequently they are observed performing the consent process until senior personnel determine that they are competent. Investigators/RAs also have weekly team meetings to discuss any difficulties that arise during consent or any other study procedure.

   Randomization: Following the baseline assessments, assessing staff will open an opaque, sealed envelop for each dyad (affected individual and caregiver). Envelops will be numbered and will contain the group assignment. A statistician not involved in the study will prepare these envelops and create a random sequence of numbers using a computer program. There will be 2 piles of envelops, one for men and one for women to recruit a similar proportions of male and female participants in both groups.
3. 1st Pilot-test Phase. Affected individual/caregiver dyads who consented will be invited to participate in the first pilot phase of 10 dyads. These subjects will participate in either Group 1 (initial intervention), which will participate first, or Group 2 (wait list control group). Group 1 will participate in the Paired PLIÉ program 2 times/week for 45 minutes for 4 weeks and then once/month for additional 3 months while Group 2 will be wait-listed. After Group 1 has completed their training, Group 2 will participate in the PLIÉ program 2 times/week for 45 minutes for 4 weeks and then once/month for additional 3 months. Group assignment will be random. Investigators will strive to have an equal distribution of men/women in the two groups.

   Intervention: the exercise protocol is based on the PLIÉ protocol, which the investigators have developed in consultation with experts worldwide who have experience performing different types of exercises in individuals with mild-to-moderate dementia, including traditional strength-building exercises, yoga, Tai Chi and Feldenkrais. Specifically, investigators have identified exercises from each of these traditions that engage the muscles most needed to maintain independence--including lower body strength (to help with getting out of bed/chair), balance (to minimize risk of falls), upper body strength (to help with lifting), fine motor exercises (to help with activities such as eating and brushing teeth), and pelvic floor exercises (to help with continence)--and have combined them into a unique integrative exercise program. These exercises are designed to be purposeful (i.e., to achieve a goal) and to build procedural ('muscle') memory. In addition, breathing and guided meditation exercises are included to promote relaxation and well-being.

   While the PLIÉ program has been tested in a senior day care setting, investigators are combining these exercises in a new way, that they can be practiced at home in dyads of affected individuals and caregivers.
4. 2nd Pilot-test Phase. In a second phase investigators will repeat the identical protocol and intervention with 10 more dyads of affected individuals and caregivers.
5. Pre- and post-intervention assessment. Investigators will perform a variety of standard measures in all participants and caregivers. The following assessments will occur at baseline and after the 3 follow-up months. They will primarily be utilized to assess feasibility and logistics of data collection procedures. Separate appointments will be made for affected individuals and caregivers to maximize the validity of data collected (e.g., to ensure that caregivers do not 'help' affected individuals with answers to questions and feel comfortable providing information about issues such as difficult behaviors or levels of stress). Affected individuals assessments will take place at the group room. The initial caregiver assessment will take place at the caregiver's home or the group room. The first line of communication for follow-up appointments will be via telephone or in person to minimize the risk of loss of privacy. At the caregiver participant's request, further communication may be conducted via mail, email, fax or text. Caregivers will be informed that these modes of communication may increase their risk of loss of privacy. Mail, email, fax and text communications will include a confidentiality statement. The minimum amount of identifying information will be included in all communications. Study forms will include unique study ID numbers only.

ELIGIBILITY:
Inclusion Criteria:

* Affected individuals: dementia diagnosis (any type, mild to moderate severity [defined as independent in at least 1 basic ADL])
* Ambulatory and able to take 2 steps without cane or walker
* Living in the community in a private home or apartment
* English language fluency.
* Caregiver/care partner: lives with affected individual
* Motivated to practice regularly (4-5 times per week) at home
* Able to answer study questions related to the affected individual's functional status, mood, behaviors, quality of life and their own feelings regarding caregiving
* English language fluency.

Exclusion Criteria:

* Affected Individuals: behavioral or physical issues that would be disruptive or dangerous to themselves or others (e.g., active psychosis, drug abuse, severe behavioral issues)
* Planning to move to a facility before the end of the study period
* Terminal illness (life expectancy < 1 year)
* Non-stable dementia medication dose
* Current participation in another research study.
* Caregiver/care partner: planning to place affected individual in an institutional setting during the study period
* Terminal illness (life expectancy < 1 year)
* Behavioral or physical issues that are disruptive or dangerous.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) from Baseline to 4 months | Baseline, post-intervention (4 months)
  We will perform a variety of standard measures in all participants and caregivers. Assessments will occur at baseline, after the 4 months of intervention, and at 8 months after follow-up of 4 months. Outcomes will primarily be utilized to assess feasibility and logistics of data collection procedures.
Change in Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-cog) from baseline to 4 months | Baseline, post-intervention (4 months)
  We will perform a variety of standard measures in all participants and caregivers. Assessments will occur at baseline, after the 4 months of intervention, and at 8 months after follow-up of 4 months. Outcomes will primarily be utilized to assess feasibility and logistics of data collection procedures.

SECONDARY OUTCOMES:
Change in Quality of Life Scale in Alzheimer's Disease (QOL-AD) from baseline to 4 months | Baseline, post-intervention (4 months)
  same as above
Change in Caregiver Burden Inventory (CBI) from baseline to 4 months | Baseline, post-intervention (4 months)
  same as above

CONTACTS AND LOCATIONS:
Overall Officials: Wolf E Mehling, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCaliforniaSF, San Francisco, California, United States

REFERENCES:
- [Background] Alzheimer's Association. 2013 Alzheimer's disease facts and figures. Alzheimers Dement. 2013 Mar;9(2):208-45. doi: 10.1016/j.jalz.2013.02.003. PMID 23507120
- [Background] Acosta D, Wortmann M. World Alzheimer Report: Alzheimer's Disease International. 2009
- [Background] Hurd MD, Martorell P, Delavande A, Mullen KJ, Langa KM. Monetary costs of dementia in the United States. N Engl J Med. 2013 Apr 4;368(14):1326-34. doi: 10.1056/NEJMsa1204629. PMID 23550670
- [Background] Rockwood K. Size of the treatment effect on cognition of cholinesterase inhibition in Alzheimer's disease. J Neurol Neurosurg Psychiatry. 2004 May;75(5):677-85. doi: 10.1136/jnnp.2003.029074. PMID 15090558
- [Background] Olazaran J, Reisberg B, Clare L, Cruz I, Pena-Casanova J, Del Ser T, Woods B, Beck C, Auer S, Lai C, Spector A, Fazio S, Bond J, Kivipelto M, Brodaty H, Rojo JM, Collins H, Teri L, Mittelman M, Orrell M, Feldman HH, Muniz R. Nonpharmacological therapies in Alzheimer's disease: a systematic review of efficacy. Dement Geriatr Cogn Disord. 2010;30(2):161-78. doi: 10.1159/000316119. Epub 2010 Sep 10. PMID 20838046
- [Background] Beeber AS, Thorpe JM, Clipp EC. Community-based service use by elders with dementia and their caregivers: a latent class analysis. Nurs Res. 2008 Sep-Oct;57(5):312-21. doi: 10.1097/01.NNR.0000313500.07475.eb. PMID 18794715
- [Background] Yao L, Giordani BJ, Algase DL, You M, Alexander NB. Fall risk-relevant functional mobility outcomes in dementia following dyadic tai chi exercise. West J Nurs Res. 2013 Mar;35(3):281-96. doi: 10.1177/0193945912443319. Epub 2012 Apr 19. PMID 22517441
- [Background] Deweer B, Ergis AM, Fossati P, Pillon B, Boller F, Agid Y, Dubois B. Explicit memory, procedural learning and lexical priming in Alzheimer's disease. Cortex. 1994 Mar;30(1):113-26. doi: 10.1016/s0010-9452(13)80327-9. PMID 8004981
- [Background] Zeller JB, Herrmann MJ, Ehlis AC, Polak T, Fallgatter AJ. Altered parietal brain oxygenation in Alzheimer's disease as assessed with near-infrared spectroscopy. Am J Geriatr Psychiatry. 2010 May;18(5):433-41. doi: 10.1097/JGP.0b013e3181c65821. PMID 20220582
- [Background] Markovich NIa, Proskuriakova AM. [Discovery of Anopheles messeae Fall. breeding sites at the Sayan reservoir and in the tailrace of the Yenisei in the construction area of Sayan-Shushenskoe hydroelectric station]. Med Parazitol (Mosk). 1986 Jan-Feb;(1):10-3. No abstract available. Russian. PMID 3959992
- [Result] Wu E, Barnes DE, Ackerman SL, Lee J, Chesney M, Mehling WE. Preventing Loss of Independence through Exercise (PLIE): qualitative analysis of a clinical trial in older adults with dementia. Aging Ment Health. 2015;19(4):353-62. doi: 10.1080/13607863.2014.935290. Epub 2014 Jul 14. PMID 25022459
- [Result] Barnes DE, Mehling W, Wu E, Yaffe K, Flores C, Chesney M. Preventing Loss of Independence through Exercise (PLIÉ): An Integrative Exercise Program for Individuals with Dementia. American Academy of Neurology; March 20, 2013, 2013; San Diego, CA
- [Result] Barnes DE, Mehling W, Wu E, Beristianos M, Yaffe K, Skultety K, Chesney MA. Preventing loss of independence through exercise (PLIE): a pilot clinical trial in older adults with dementia. PLoS One. 2015 Feb 11;10(2):e0113367. doi: 10.1371/journal.pone.0113367. eCollection 2015. PMID 25671576